CLINICAL TRIAL: NCT05852808
Title: Evaluation of Pain Level Reduction After Low-dose Radiation in Symptomatic Facet Joint Arthritis - A Prospective Randomized Clinical Trial.
Brief Title: Evaluation of Pain Level Reduction After Low-dose Radiation in Symptomatic Facet Joint Arthritis
Acronym: LORAFA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: bad recruiting
Sponsor: Silvia Gomez Ordonez (Other)
Responsible Party: Sponsor-Investigator, Silvia Gomez Ordonez, Dr. med., Kantonsspital Aarau
Organization: Kantonsspital Aarau (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-00272; ex22Gomez
Record Dates: First submitted 2023-04-28; First posted 2023-05-10 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Lower Back Pain Chronic; Facet Joint Arthrosis; Osteoarthritis, Spine
Keywords: Low dose radiation therapy; SPECT-CT; facet joint steroid injection
MeSH Terms: conditions — Osteoarthritis, Spine | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Prospective non-inferiority double-arm randomized controlled single centre trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-articular steroid injections (Active Comparator): The intra-articular steroid injections are the most common standard of care to treat the lower back pain resulting from FJA.
  Interventions: Drug: Intra-articular steroid injections
- Low-dose radiation therapy (Experimental): LDRT is commonly used as treatment for benign degenerative inflammatory disorders
  Interventions: Radiation: Low-dose radiation therapy

INTERVENTIONS:
Drug: Intra-articular steroid injections — The patient will be placed in prone position and the facet joints will be imaged by pa-radiation path with attention to radiation protection. 20 mg Kenacort + 1 ml Bupivacain (2.5 mg/ml) will be injected into the affected facet joints. The patient is monitored after the intervention for another 30 minutes before leaving the hospital. In order to track the pain level, the patient will be instructed to keep a pain diary. The patient will be contacted via telephone 72h after the intervention and asked about the pain level.
  The intervention is finished after one consultation.
  Arms: Intra-articular steroid injections
Radiation: Low-dose radiation therapy — The treatment consists of an informing consultation, a planning CT scan and a series of 10 radiation sessions delivered over 3.5 weeks ( = 12 visits in total). The clinical target volume (CTV) will be defined based on the MRI and SPECT/CT. Planning target volume (PTV) will be expanded in all directions by 0.5 cm beyond the CTV. Patients will be treated in a supine position with minimum 6 MV photons and a 3D-technique or volumetric modulated arc therapy (VMAT)-technique. A kilovolt (kV) and in exception a cone-beam CT will be performed before each treatment for positioning accuracy. A dose of 0.5 Gy x 10 fractions (3 times per week) will be delivered over 3.5 weeks. Each radiotherapy treatment session takes approximately 15 minutes. If a second radiotherapy series will be done (NRS 4-10 at visit 4), the radiotherapy dose und fractionation will be the same as the first series.
  Arms: Low-dose radiation therapy

SUMMARY:
The goal of this clinical trial is to compare low-dose radiation therapy (LDRT) with intra-articular steroid injections in participants suffering from chronic lower back pain as cause of facet joint arthritis (FJA).

The main question[s] it aims to answer are:

* Is LDRT non-inferior to intra-articular steroid injections in terms of pain reduction
* Is there a difference in long-term pain reduction between LDRT and intra-articular steroid injections Participants will be randomly assigned to one of the two treatment groups.

DETAILED DESCRIPTION:
However, there has been no published study providing scientific evidence by prospective randomized data on the effect of LDRT in patient suffering from facet osteoarthritis. LDRT seems a viable treatment method with anti-inflammatory potential and possible long-lasting benefit in pain resolution for patients with facet joint arthritis (FJA), which can prevent from an ultimate surgical treatment.

The rationale of this trial is to generate scientific evidence that LDRT is an alternative non-invasive treatment option for FJA, whose primary outcome "pain reduction" is equivalent to the most common treatment intra-articular steroid injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative symptomatic facet joint osteoarthritis confirmed by MRI (lumbar spine) and standing X-ray
* Patients who underwent treatment for facet joint syndrome at the Dept. of Orthopaedic Surgery and Traumatology of KSA (Kantonsspital Aarau) or Dept. of Rheumatology of KSA or Dept. of Neurosurgery of KSA, onset of symptoms and treatment with pain medication and physiotherapy
* The informed consent form for participation in the study was signed
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Age ≥ 45 years
* Karnofsky Performance Status (KPS) ≥ 80 %
* Ability to take steroids and bridge or pause NOAC (New oral anticoagulants) / Marcoumar
* Show a positive Tracer-Uptake in the SPECT-CT in max. 4 facet joints of the lumbar spine (regardless of radiologic changes in MRI or CT)
* Immediate ≥ 70% pain reduction after 1 positive diagnostic infiltration of the suspected facet joint(s)
* Negative middle-/long-term effect (4-12 weeks after first steroid injection, defined as "NRS 5-10 at 4-12 weeks")

Exclusion Criteria:

* Any previous infiltration therapy in the suspected spine region (+/- 3 segments) within the last 3 years
* Any previous radiotherapy, radiofrequency ablation, other pain modulating interventions (e.g. thermos/-cryoablation or spinal cord stimulators) or surgery in the suspected spine region (+/- 3 segments)
* Prior or concurrent malignancy (≤ 5 years prior to enrolment in study) except: nonmelanoma skin cancer, cervix carcinoma in situ, prostatic intraepithelial neoplasia) Contraindications to radiotherapy (for example connective tissue disorders such as scleroderma)
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Pregnancy, desire to have own children or lactation during study participation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Change in pain level, measured on a numeric rating scale (NRS) | Baseline and 3 month after randomization
  Difference in pain score on a numeric rating scale (NRS) with values from 0 to 10 (0 = no pain, 10 = highest imaginable pain)

SECONDARY OUTCOMES:
Number of reported (serious) adverse events ((S)AE) | Up to 12 months
  Toxicity of LDRT measured by number and description of reported (S)AE (serious adverse events)
Percentage of patients with NRS<4 (equals responders) after first treatment session | Up to 3.5 weeks
  Efficacy of LDRT measured by percentage of patients with NRS<4 (equals responders) after first treatment session.
Percentage of patients with NRS<4 (equals responders) after six months | At six months
  Efficacy of LDRT measured by percentage of patients with NRS<4
Change in pain level, measured on a numeric rating scale (NRS) | Baseline, at 6 and 12 months after randomization
  Difference in pain score on a numeric rating scale (NRS) with values from 0 to 10 (0 = no pain, 10 = highest imaginable pain)
Change in quality of life measured by the Short Form Health (SF)-36 questionnaire | Baseline, at 3, 6 and 12 months after randomization
  The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health or emotional wellbeing

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Gomez Ordonez, Dr. med., Principal Investigator — Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Switzerland